CLINICAL TRIAL: NCT04090762
Title: Improving Perinatal Outcomes Using Conditional and Targeted Transfers
Acronym: IMPACTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Principal Investigator, Edward Okeke, Senior Economist, RAND
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01HD090231 (NIH)
Record Dates: First submitted 2019-06-28; First posted 2019-09-16 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Utilization, Health Care; Birth Outcomes
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Women in the control arm will complete the baseline and follow up surveys but will not receive any intervention.
- Risk information only (Active Comparator): Women in the risk only arm who exhibit characteristics associated with a greater risk of a poor birth outcome will be informed that they possess these characteristics. Risk characteristics (identified from the medical and epidemiological literature) include age, prior pregnancy and birth history (e.g., previous stillbirth).
  Interventions: Behavioral: Risk information provision
- Conditional Cash Transfer only (Active Comparator): Women in this arm will be eligible to receive conditional cash transfers. To receive the transfer, pregnant women must attend prenatal care and give birth in a health facility.
  Interventions: Behavioral: Conditional cash transfer
- Conditional Cash Transfer and risk information (Active Comparator): Women in this arm will be provided with risk information at the time of baseline survey administration AND be eligible to receive conditional cash transfers, pending attendance at prenatal care and delivery at a health facility.
  Interventions: Behavioral: Conditional cash transfer; Behavioral: Risk information provision

INTERVENTIONS:
Behavioral: Conditional cash transfer — Pregnant women receive cash payments conditioned on their use of prenatal services and use of a health facility for child birth.
  Arms: Conditional Cash Transfer and risk information; Conditional Cash Transfer only
Behavioral: Risk information provision — Pregnant women who exhibit characteristics associated with a greater risk of a poor birth outcome - these will be identified from the medical and epidemiological literature - will be informed that they possess these characteristics.
  Arms: Conditional Cash Transfer and risk information; Risk information only

SUMMARY:
It has been estimated that increasing the use of skilled care during childbirth could prevent up to 1.5 million maternal and newborn deaths and stillbirths by 2025. Conditional cash transfer programs, in which women receive cash payments conditioned on the use of maternal health services, are increasingly being used as a mechanism to increase uptake. In this study, the investigators randomly assign households to receive varying cash amounts conditioned on uptake of recommended pregnancy and delivery care. The investigators crosscut this with an intervention in which pregnant women receive information about their risk type. This randomized trial will provide new evidence about the potential efficacy of targeting cash transfers by pregnancy risk. This study will take place in 288 primary health service areas (HSAs) in Nigeria.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ages 15-49 who reside in the participating health service areas

Exclusion Criteria:

* none

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36607 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Probability of prenatal care | 3-4 months after anticipated childbirth/delivery date
  the probability of receiving prenatal care
Uptake of prenatal care | 3-4 months after anticipated childbirth/delivery date
  the number of prenatal visits completed
Uptake of health facility birth | 3-4 months after anticipated childbirth/delivery date
  probability of giving birth at a health facility
Child mortality - fetal loss | 3-4 months after anticipated childbirth/delivery date
  Child mortality - fetal loss
Child mortality - stillbirths | 3-4 months after anticipated childbirth/delivery date
  Child mortality - stillbirths
Child mortality - early infant death | 3-4 months after anticipated childbirth/delivery date
  Child mortality - early infant death

SECONDARY OUTCOMES:
Maternal health | 3-4 months after anticipated childbirth/delivery date
  delivery complications
Maternal mortality | 3-4 months after anticipated childbirth/delivery date
  maternal death
Child weight | 3-4 months after anticipated childbirth/delivery date
  Child weight
Child length | 3-4 months after anticipated childbirth/delivery date
  Child length
Uptake of postnatal care | 3-4 months after anticipated childbirth/delivery date
  Probability of using postnatal care
Child vaccination | 3-4 months after anticipated childbirth/delivery date
  Probability of receiving recommended child immunizations
Maternal beliefs | 3-4 months after anticipated childbirth/delivery date
  Risk perceptions and beliefs assessed using a questionnaire
Pregnancy behavior - tetanus vaccination | 3-4 months after anticipated childbirth/delivery date
  Probability of receiving tetanus vaccination
Pregnancy behavior - malaria prophylaxis | 3-4 months after anticipated childbirth/delivery date
  Probability of receiving malaria prophylaxis
Pregnancy behavior - blood building products | 3-4 months after anticipated childbirth/delivery date
  Probability of receiving blood building products
Pregnancy behavior - dietary consumption | 3-4 months after anticipated childbirth/delivery date
  Probability of consuming nutrient-rich foods assessed using questionnaire
Quality of perinatal care | 3-4 months after anticipated childbirth/delivery date
  Quality score assessed using a questionnaire
Timely initiation of prenatal care | 3-4 months after anticipated childbirth/delivery date
  Probability of initiating prenatal care in the first trimester of pregnancy
Maternal work | 3-4 months after enrollment
  Hours worked in the last seven days

OTHER OUTCOMES:
Maternal depression | 3-4 months after anticipated childbirth/delivery date
  Depression assessed using the Edinburgh Postnatal Depression Scale
Health facility choice | 3-4 months after anticipated childbirth/delivery date
  Probability of receiving care at a government or private hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Aminu Kano Teaching Hospital, Kano, Kano State, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okeke EN, Abubakar IS, De Guttry R. In Nigeria, Stillbirths And Newborn Deaths Increased During The COVID-19 Pandemic. Health Aff (Millwood). 2021 Nov;40(11):1797-1805. doi: 10.1377/hlthaff.2021.00659. Epub 2021 Oct 20. PMID 34669501
- [Background] Okeke EN. Playing defense? Health care in the era of Covid. J Health Econ. 2022 Sep;85:102665. doi: 10.1016/j.jhealeco.2022.102665. Epub 2022 Jul 25. PMID 35952443